CLINICAL TRIAL: NCT02115659
Title: Randomized Controlled Trial of Triptolide-Containing Formulation for Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Triptolide-Containing Formulation as Treatment for Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Mei changlin, Professor,Director of the Kidney Institute, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CZKIPLA-ADPKD-002
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD; triptolide
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo plus standard treatment. Anti-hypertension drug(s) for hypertension; Antibiotics for cyst infections; cause oriented treatment for flank pain.
  Interventions: Drug: Placebo
- Triptolide-Containing Formulation (Experimental): Triptolide-Containing Formulation (1mg/kg/d) was prescribed; Dosage will be adjusted if necessary according to the adverse events monitoring.
  Interventions: Drug: Triptolide-Containing Formulation

INTERVENTIONS:
Drug: Triptolide-Containing Formulation — Triptolide-Containing Formulation (1mg/kg/d) plus standard treatment of complications. Anti-hypertension drug(s) for hypertension; Antibiotics for cyst infections; cause oriented treatment for flank pain.
  Other Names: Triptolide-Containing Formulation plus standard treatment.
  Arms: Triptolide-Containing Formulation
Drug: Placebo — Placebo plus standard treatment of complications. Anti-hypertension drug(s) for hypertension; Antibiotics for cyst infections; cause oriented treatment for flank pain, etc.
  Other Names: Placebo plus standard treatment.
  Arms: Placebo

SUMMARY:
Triptolide was shown in experimental studies to inhibit the cyst formation and growth in ADPKD models, while triptolide-containing formulation was revealed to potentially slow the disease progression in several proteinuric ADPKD patients in our clinical practice. It remains to be shown the effect of triptolide-containing formulation on total kidney volume (TKV) enlargement and renal function protection in ADPKD patients.

DETAILED DESCRIPTION:
Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patient older then 40 years of age without gender limitation
* Estimated glomerular filtration rate (eGFR) higher than 60 ml/min 1.73m2
* documented kidney volume progression with yearly increasing rate more than 6%
* informed consent

Exclusion Criteria:

* Female who is planning to become pregnant, who is pregnant and/or lactating, who is unwilling to use effective means of contraception
* impaired liver function as increased liver enzymes (2-fold above normal values)
* uncontrolled hypercholesterolemia (fasting cholesterol > 8 mmol/l) or hypertriglyceridaemia (> 5 mmol/l) under lipid lowering therapy
* granulocytopenia (white blood cell < 3,000/mm3) or thrombocytopenia (platelets < 100,000/mm3)
* hepatitis B or C, HIV infection
* malignancy
* mental illness that interfere with the patient ability to comply with the protocol
* drug or alcohol abuse
* known hypersensitivity to similar drugs as Triptolide-Containing Formulation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
renal volume measured by high resolution magnetic resolution imaging | 2 yrs

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | 2 yrs
Adverse events. | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China